CLINICAL TRIAL: NCT03257917
Title: Understanding Out-of-pocket Expenses and Patient Time Spent on Healthcare in Metastatic Breast Cancer Patients (Understanding Value in Metastatic Breast Cancer)
Brief Title: Understanding Value in Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Gabrielle Rocque, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-170504005
Record Dates: First submitted 2017-07-26; First posted 2017-08-22 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Metastatic Breast Cancer
Keywords: Financial Burden; Out of Pocket expenses; Time spent on Healthcare; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Understanding value in Metastatic Breast Cancer — The overall objective of this project is to gain knowledge about out-of-pocket (OOP) expenses and lost opportunity costs among metastatic breast cancer (MBC) patients. To achieve this objective, MBC patients will be asked to participate in a short, 37-question survey asking questions about the financial burden, OOP expenses, and opportunity costs related to their cancer care.

SUMMARY:
The overall objective of this project is to gain knowledge about out-of-pocket (OOP) expenses and lost opportunity costs among metastatic breast cancer (MBC) patients. To achieve this objective, MBC patients will be asked to participate in a short, 37-question survey asking questions about the financial burden, OOP expenses, and opportunity costs related to their cancer care

DETAILED DESCRIPTION:
The treating physician, PI or study coordinator will inform eligible MBC patients about the study via a letter (Appendix B) during or prior to their regular clinic visits in a waiting area. Prior to the survey administration, study coordinator will obtain all necessary signatures on the ICF from interested study participants in the private clinic room or infusion area. The survey (Appendix A) will consist of 37 survey questions, which should take patients less than 30 minutes to complete during their regularly scheduled clinic visit. Study participants will have the option of taking incomplete surveys home, completing, and mailing it back to us using stamped, self-addressed envelopes provided during their clinic visit. All consented participants will also be given the option to complete the survey over the phone with a study coordinator. Participants will be requested to provide their preferable times and days for a phone call with a coordinator. The study coordinator will call the patient and administer the same survey that would be given during a clinic visit. If participants prefer completing the survey in the clinic a research coordinator will remain in the room and will verbally facilitate the completion of the survey. Participants will be compensated in the form of merchandise at the time they agree to participate (the photo of sample merchandise is attached). Surveys will be collected by the study coordinator and stored in secure, locked rooms at the UAB Comprehensive Cancer Center, where the study coordinators will double-key enter de-identified survey responses into an encrypted, password protected, electronic database.

ELIGIBILITY:
Inclusion Criteria:

* All female MBC patients 18 years of age and older who have received treatment within the past two years at UAB

Exclusion Criteria:

* Non-English speakers, patients residing in nursing homes or receiving hospice care

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The participants will be derived from Metastatic Breast Cancer patients receiving care at UAB Kirklin Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Post-cancer diagnosis cost | 2 years
  based on a validated survey

SECONDARY OUTCOMES:
Time loss experienced by patients with metastatic breast cancer. | 2 years
  based on a validated survey
Do patient characteristics (sociodemographics, cancer characteristics, health status, healthcare utilization) influence the total cost of care or financial burden? | 2 Years
Does treatment type (chemotherapy vs. hormone therapy) influence the total cost of care or financial burden? | 2 years
What is the trajectory of financial burden or total cost of care over time (year pre-MBC diagnosis vs. post-MBC diagnosis)? | 2 Years
Does financial burden or total cost of care influence treatment adherence? | 2 years
Does clinical trial participation influence the total cost of care or financial burden? | 2 years
Does financial burden or total cost of care influence perception of or preference for shared decision-making? | 2 years
Describe the cost experienced by patients with metastatic breast cancer. | 2 years
Describe the productivity loss experienced by patients with metastatic breast cancer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle B Rocque, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No